CLINICAL TRIAL: NCT00363506
Title: Nutritional Based Protocol to Balance Serotonin for the Prevention or Reduced Frequency/Duration/Intensity of Migraines
Brief Title: American Migraine Prevention Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dynamic Health Resources (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DHR-757962-7081
Record Dates: First submitted 2006-08-09; First posted 2006-08-15 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Migraine Disorders
Keywords: nutritional; C10.228.140.546.399.750
MeSH Terms: conditions — Migraine Disorders

INTERVENTIONS:
Behavioral: Serotona Plus and dietary behavior management

SUMMARY:
The purpose of this study is to evaluate the use of nutritional supplementation and dietary management for the reduction in frequency, duration, and intensity of migraine headache pain.

DETAILED DESCRIPTION:
AMPS, the American Migraine Prevention Study Program is a home based nutritional study for migraine prevention. It is designed to evaluate a nutritional supplement along with proper diet, and trigger management that may prevent migraines or reduce the frequency, duration and intensity of migraine headache pain.

The AMPS Program is availalbe nationwide. It is a home based study program.

During the three month study period, participants will be asked to take a daily nutritional supplement and follow a recommended diet to avoid potential migraine triggers. Participants will be asked to maintain a headache log and submit headache questionnaires at the beginning and end of the study. Participants do not have to travel and can participate from their current location.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of migraines
* Ages 18-72
* Migraines more than once per month
* Diagnosed migraines for more than one year

Exclusion Criteria:

* Pregnant/nursing

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-01; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Migraine Impact and Disability Survey (MIDAS) - symptoms measured at study beginning and at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: John J Carvalho, MBA, Study Chair — Dynamic Health Resources
Locations (1):
- Nationwide home based study program, Chesapeake, Virginia, United States